CLINICAL TRIAL: NCT00147797
Title: Influence of Pravastatin on Carotid Artery Structure and Function in HIV-infected Patients Under Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: Saint Antoine University Hospital (Other)
Collaborators: French Cardiology Society (Other)
Other Study IDs: 2003-01; 53-03
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2007-04

CONDITIONS: HIV Infection; Carotid Atherosclerosis; Dyslipidemia
Keywords: Atherosclerosis; intima media thickness; aortic stiffness; HIV infection; Dyslipidemia; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Carotid Artery Diseases; Dyslipidemias; Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- Pravastatin group: Patients in the pravastatin group were consecutively recruited in four department of infectious diseases if they fulfilled the following criteria : (1) HIV-infected treated with HAART for > 12 months 2) with dyslipidemia, defined as fasting serum LDL cholesterol > 160 mg/dL before initiation of pravastatin, (3) treated with pravastatin > 12 months and one more coronary risk factor.
- COotrol group: The patients in the control group were selected consecutively in the same departments among 1) HIV-infected patients treated with HAART > 12 months 2) fasting serum LDL cholesterol > 160 mg/dL 3) without lipid-lowering drugs and one more coronary risk factor. Cases and control patients were matched for age, gender and tobacco consumption.

SUMMARY:
The advent of new antiretroviral agents, in particular Highly Active Antiretroviral Therapy (HAART), spectacularly reduced HIV-associated morbidity and mortality. However, new complications have appeared in HIV-infected patients treated by with HAART such as dyslipidemia, insulin resistance, diabetes mellitus, and related cardiovascular complications including acute coronary syndromes, peripheral vascular disease, and stroke have been reported.

A linear association has been proved between increased intima-media thickness of the common carotid artery (CCA-IMT), aortic stiffness (pulse wave velocity [aPWV]) and incidence of cardiovascular events suggesting that IMT and aPWV could be considered as an early marker of atherosclerosis. The progression of IMT has been shown to be predictive of cardiovascular events. Case control and longitudinal studies but not all have suggested an increase CCA-IMT in HIV-infected patients under HAART compared with non-HIV infected patients with different progression.

The aim of this study was to examine the effects of pravastatin on CCA-IMT and aortic stiffness in dyslipidemic HIV-infected patients receiving HAART by using a high-resolution echotracking system.

Patients in the pravastatin group were consecutively recruited in four department of infectious diseases if they fulfilled the following criteria : (1) HIV-infected treated with HAART for > 12 months 2) with dyslipidemia, defined as fasting serum LDL cholesterol > 160 mg/dL before initiation of pravastatin, (3) treated with pravastatin > 12 months and one more coronary risk factor. The patients in the control group were selected consecutively in the same departments among 1) HIV-infected patients treated with HAART > 12 months 2) fasting serum LDL cholesterol > 160 mg/dL 3) without lipid-lowering drugs and one more coronary risk factor. Cases and control patients were matched for age, gender and tobacco consumption.

Using data from Mercie et al., inclusion of 42 patients in pravastatin and control groups was the minimum sample size needed for detection of a 6.5% difference in CCA-IMT, in a two-sided test (a = 0.05, b = 0.20).

The protocol of the study, sponsored by the French Society of Cardiology was approved by the Committee for the Protection of Human Subjects in Biomedical Research of Pitié-Salpétrière University hospital in Paris. Written informed consent to participate in the study was obtained from each patient.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients treated with HAART for > 12 months
* With dyslipidemia, defined as LDL cholesterol > 160 mg/dL before initiation of statin
* Treated with pravastatin > 12 months and one more coronary risk factor. The patients in the control group were selected consecutively in the same departments among

  * HIV-infected patients treated with HAART > 12 months
  * LDL cholesterol > 160 mg/dL
  * Without lipid-lowering drugs and one more coronary risk factor. Cases and control patients were matched for age, gender and tobacco consumption.

Exclusion Criteria:

* Patients with history of coronary artery disease, peripheral artery disease, endarterectomy, aortic dissection

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2003-05; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Laurent, MD, PhD, Study Director — Department of Pharmacology and INSERM U652, Hôpital Européen Georges Pompidou, Paris, France
Locations (1):
- Department of Pharmacology and INSERM U652, Hôpital Européen Georges Pompidou, Paris, France